CLINICAL TRIAL: NCT05517044
Title: The PRe-Acclimatization auGmented extreMe Altitude eXpedition (PRAGMAX) Randomized Controlled Trial
Brief Title: The Pre-acclimatization Augmented Extreme Altitude Expedition
Acronym: PRAGMAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss Sportclinic Bern (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BASEC 2022-00679
Record Dates: First submitted 2022-08-03; First posted 2022-08-26 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Altitude Hypoxia; Perfusion; Complications
Keywords: Microcirculation; Oxygen delivery capacity; Preacclimatization; nitrogen concentration tent
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Two independent randomized-controlled trials with each an intervention and a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preacclimatization group (Experimental): The participants assigned to the preacclimatization group will undergo a defined preacclimatization program by sleeping in a nitrogen concentration tent prior to an expedition to high altitude.
  Interventions: Other: Nitrogen tent preacclimatization to high altitude
- Control group (No Intervention): The participants assigned to the control group sleep in their regular environment without use of a nitrogen concentration tent prior to an expedition to a high altitude expedition.

INTERVENTIONS:
Other: Nitrogen tent preacclimatization to high altitude — The participants assigned to the preacclimatization group spend a minimum of six hours during sleep, throughout the acclimatization period (four weeks preceding the expedition) in a nitrogen concentration tent (Hypoxico OHG, Traunstein, Germany) set to an environmental PO2 corresponding to an altitude of 2500 masl, with a progression to 5500 masl within 28 days in steps of 1000 m every seven days. Respiratory Polygraphy is used to detect periodic breathing, SpO2, and heart rate continuously during sleep and is performed before and after the designated preacclimatization period, and repetitively when increasing normobaric hypoxia in the group with nitrogen concentration tent preacclimatization.
  Arms: Preacclimatization group

SUMMARY:
The aim of this study is to investigate the effect of pre-acclimatization in a nitrogen tent at home, ventilated with a slightly increased nitrogen percentage, in preparation for an expedition at extreme altitude. Specifically, the current study aims to gather knowledge, whether pre-acclimatization, first, leads to improved capillary function during an expedition to extreme altitude, and second, affects incidence of altitude sickness and the likelihood of reaching the expedition destination without oxygen supplementation.

The project will be carried out in two phases corresponding to two randomized controlled trials in healthy volunteers, who are participating in an expedition at extreme altitudes with or without pre-acclimatization.

DETAILED DESCRIPTION:
Expeditions to the world's highest peaks are attempted by increasing numbers of alpinists, taking advantage of broad commercial support. At extreme altitude successful functioning, and even survival, are only possible with adequate acclimatization, which consists of time-consuming exposure to gradually higher sleeping altitudes. Generally, an increase in 300-600 m per day at altitudes above 3000 m, and the minimization of cumulative time spend above 6500 m, are considered safe practice. Mainly in an attempt to accelerate expeditions to extreme altitudes, a preacclimatization technique using nitrogen concentration tent induced normobaric hypoxia is increasingly employed in practice, and already part commercial expedition plans. Some previous research indicates that intermittent normobaric hypoxia may reduce the incidence of acute mountain sickness, while the results from other studies remain inconclusive or negative. One study has not found serious adverse effects related to intermittent normobaric hypoxia, such as high-altitude pulmonary or cerebral edema.

Thus, despite the emergence of increasing numbers of commercial expedition programs making use of nitrogen concentration tent preacclimatization protocols, many factors remain unclear. Next to remaining uncertainties regarding the extent of the hypoxic condition induced by these devices, current data does not allow adequate conclusions regarding the choice of optimal preacclimatization protocol, optimal associated ascent profiles, and possible effects on oxygen delivery capacity to the tissue, incidence of high-altitude related disease, and even summit success. Thus, the present study aims to conduct a randomized controlled trial to assess the efficacy of nitrogen concentration tent preacclimatization as part of two expeditions to extreme altitude. The immediate effects of nitrogen concentration tent preacclimatization are assessed through continuous monitoring of oxygen partial pressure in the tent and the hemoglobin oxygen saturation throughout preacclimatization. To test whether preacclimatization is associated with physiologic adaptation, tissue red blood cell perfusion as a main contributor to increase oxygen delivery capacity in the microcirculation throughout acclimatization to extreme altitude, is assessed using non-invasive handheld vital microscopy during preacclimatization and throughout the expedition, and the incidence and severity of high-altitude related disease and summit success, are recorded during the expeditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Active alpinists (active alpinists denotes individuals with regular experience in alpine high mountain climbing in rock, ice and snow terrain of difficulty WS - ZS according to the Swiss Alpine Club (SAC-CAS) grading scale assessed in a self-reporting questionnaire
* age > 18 years

Exclusion Criteria:

* history of high-altitude pulmonary edema or cerebral edema
* pregnancy or lactation
* heart failure (AHA Stage B and above)
* pulmonary hypertension
* pulmonary disease excluding mild bronchial asthma
* chronic kidney failure (KDIGO Stage 1 and above)
* chronic liver disease
* subjects with a history of smoking (> 5 PY), and high familiar predisposition for cardiovascular disease, when combined with smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difference in sublingual total capillary vessel density (TVD) induced by preacclimatization and high-altitude exposure (change from baseline) | Microcirculation assessment taken: 4 and 1 week prior to the expedition start (preacclimatization), Day 5 to 10 of the expedition in Nepal, Day 2 after the return from Nepa
  Sublingual microcirculatory functional hemodynamic variable measured using a handheld vital microscopy. (ref: Communications Biology 2019; 2: 217 UND ref. Curr Opin Crit Care 2020; 26: 273-280.)
Difference in sublingual functional capillary density (FCD) induced by preacclimatization and high-altitude exposure (change from baseline) | Microcirculation assessment taken: 4 and 1 week prior to the expedition start (preacclimatization), Day 5 to 10 of the expedition in Nepal, Day 2 after the return from Nepa
  Sublingual microcirculatory functional hemodynamic variable measured using a handheld vital microscopy. (ref: Communications Biology 2019; 2: 217 UND ref. Curr Opin Crit Care 2020; 26: 273-280.)
Difference in sublingual red blood cell velocity (RBCv) induced by preacclimatization and high-altitude exposure (change from baseline) | Microcirculation assessment taken: 4 and 1 week prior to the expedition start (preacclimatization), Day 5 to 10 of the expedition in Nepal, Day 2 after the return from Nepa
  Sublingual microcirculatory functional hemodynamic variable measured using a handheld vital microscopy. (ref: Communications Biology 2019; 2: 217 UND ref. Curr Opin Crit Care 2020; 26: 273-280.)
Difference in sublingual capillary hematocrits (cHct) induced by preacclimatization and high-altitude exposure (change from baseline) | Microcirculation assessment taken: 4 and 1 week prior to the expedition start (preacclimatization), Day 5 to 10 of the expedition in Nepal, Day 2 after the return from Nepa
  Sublingual microcirculatory functional hemodynamic variable measured using a handheld vital microscopy. (ref: Communications Biology 2019; 2: 217 UND ref. Curr Opin Crit Care 2020; 26: 273-280.)
Difference in sublingual Tissue red blood cell perfusion (tRBCp) induced by preacclimatization and high-altitude exposure (change from baseline) | Microcirculation assessment taken: 4 and 1 week prior to the expedition start (preacclimatization), Day 5 to 10 of the expedition in Nepal, Day 2 after the return from Nepa
  Sublingual microcirculatory functional hemodynamic variable measured using a handheld vital microscopy. (ref: Communications Biology 2019; 2: 217 UND ref. Curr Opin Crit Care 2020; 26: 273-280.)

SECONDARY OUTCOMES:
Change in acute mountain sickness (Lake Louise score) | LLS_AMS score reported: 4 and 1 week prior to the expedition start (preacclimatization), Day 5 to 10 of the expedition in Nepal, Day 2 after the return from Nepal
  Efficacy of the nitrogen concentration tent for high altitude preacclimatization by means of incidence and severity of acute mountain sickness (LLS-AMS score)
Summit success | Day 9 of the expedition in Nepal (Summit attempt)
  Efficacy of nitrogen concentration tent for high altiude preacclimatization by means of incidence and severity of summit success
Nitrogen tent | 4 weeks (prior to the expedition start (preacclimatization))
  Proportion of preacclimatization time in the nitrogen concentration tent within the target environmental oxygen partial pressure within a 5% boundary
Low hemoglobin oxygen saturation | 4 weeks (prior to the expedition start (preacclimatization))
  Proportion of preacclimatization time with a hemoglobin oxygen saturation below 90%
Hemoglobin oxgen saturation dips | 4 weeks (prior to the expedition start (preacclimatization))
  Occurrence of dips in hemoglobin oxygen saturation below 80% for >5 min during preacclimatization

CONTACTS AND LOCATIONS:
Overall Officials: Matthias P Hilty, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No